CLINICAL TRIAL: NCT06888206
Title: Impact of Age on Mortality in Critically Ill Adult Patients in Nepal- a Single Center Retrospective Study of 5 Years.
Status: Completed | Type: Observational
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Bipin Karki, Principle Investigator, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Other Study IDs: 400(6-11)E2- 081/082
Record Dates: First submitted 2025-03-15; First posted 2025-03-21 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Effect of Age on Mortality; ICU Mortality; Age
Keywords: Age; Mortality; Intensive care unit; Low-middle income country

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Young adult: Patients admitted to the ICU in the age group less than 24
- Adult: Adults of the age group 25-44
- Middle age: Patients of the age group 45-64
- Older adult: Patients of the age group >65 years

SUMMARY:
Rationale: Age is often considered a strong factor that determines the outcomes in critically ill patients. In a resource limited low middle income country (LMIC) like Nepal, the age factor is often considered when making treatment decisions by family especially when considering limiting treatment modalities. Whether or not this consideration of age for outcome prediction is appropriate however is a different discussion especially considering the fact that actual data from Nepalese ICUs are missing.

Study Objective: To find the impact of age on mortality in critically ill patients.

Design: A registry based, retrospective, descriptive study. Sample size: Convenience sampling of all the patients who are admitted to the ICU.

Duration: Retrospective data from the 5-year period between November, 2019 to December, 2024.

Place: Intensive care units (ICUs), Tribhuvan University Teaching Hospital (TUTH).

Interventions: Not applicable Expected results: The study will help determine the mortality of the critically ill adult patients in terms of age.

DETAILED DESCRIPTION:
Age is often considered a poor prognostic factor for most disease conditions. However the effect of age on mortality may not be as simple. Few studies have shown contradicting results such that chronological age exerted no effect on mortality. This may be due to the effect of physiological reserve and well being more than the chronological age.

It has to be noted that with improvement in the overall health care along with the increase in the average life expectancy, ICUs all over the world will be facing a lot more of an "aged" population.

This is even more relevant in our context. The average life expectancy at birth in Nepal has significantly gone up from about 65 years in 2000 AD to 70 years in 2021. This can be expected to improve further with improvements in neonatal and child mortality rates, immunization rates, the health care system delivery and reach. With this, the adult care medicine in Nepal should gear up to face older patients with a new set of challenges including increasing frailty, increasing comorbidities, increased requirements of supportive therapy including rehabilitation and nutrition.

As of now age is often considered a significant factor for making health decisions in Nepal. In a resource limited setting in such an LMICs where a majority of the population lack health insurance coverage, health care costs are borne by the family.

This, when added to the general notion that elderly patients have a poor prognosis, may lead to an unfounded decision to limit treatment decisions including withdrawal of treatments from the ICU.

Rationale and Justification of study This study will help to determine the age related mortality of patients admitted to the ICU. As per the knowledge of the authors, no such large scale studies have been published from Nepal.

ELIGIBILITY:
Inclusion Criteria:

Age>18 years Admission to the ICU

Exclusion Criteria:

None

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted to the ICUs of Tribhuvan University Teaching Hospital will be enrolled for this registry based retrospective study
Sampling Method: Non-Probability Sample
Enrollment: 8189 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
All cause ICU mortality | 2019, November to 2024 December
  * To determine the all cause ICU mortality among rates among patients in ICU grouped according to Medical Subject Heading(MeSH)
    * Young adult: 19-24 years
    * Adult: 25-44 years
    * Middle aged: 45-64 years
    * Older adult (Senior): >65 years
  * To determine the all cause ICU mortality among rates among patients in ICU grouped into decades
  * To determine the all cause ICU mortality among rates among patients >65 years in ICU according to WHO classification of elderly
    * Young-old: 60-74 years
    * Old-old: 75- 84 years
    * Oldest-Old: >85 years

CONTACTS AND LOCATIONS:
Locations (1):
- Tribhuvan University Teaching Hospital, Mahārājgañj, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Yes
The de-identified patient data may be shared with the statistician for statistical analysis
Supporting Information: Study Protocol, SAP, CSR
Time Frame: March 2025- December 2025
Access Criteria: All the de-identified patient data from the registry will be available to data handlers who will enter it in a format suitable for statistical analysis which will be available for the statistician for analysis.